CLINICAL TRIAL: NCT04804670
Title: To Determine the Effectiveness of a Sonic Toothbrush and Interdental Device With Different Toothbrush Designs to Brushing and Flossing on Plaque, Gingival Bleeding and Inflammation: a 4-week Randomized Controlled Trial
Brief Title: To Compare the Effectiveness of Three Self-care Oral Hygiene Regimens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Water Pik, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 28SFTBF2020
Record Dates: First submitted 2020-11-17; First posted 2021-03-18 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2020-11

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Sonic-Floss toothbrush and small brush head (Experimental): sonic toothbrush used for 2 minutes and water flosser used for 1 minute
  Interventions: Device: Power device A
- Sonic-Floss toothbrush and full size brush head (Experimental): sonic toothbrush used for 2 minutes and water flosser used for 1 minute
  Interventions: Device: Power device B
- Manual brushing and flossing (Active Comparator): American Dental Association standard manual toothbrush used for 2 minutes and dental floss all teeth
  Interventions: Device: Routine Oral Hygiene

INTERVENTIONS:
Device: Power device A — Oral hygiene regimen completed daily
  Arms: Sonic-Floss toothbrush and small brush head
Device: Power device B — Oral hygiene regimen completed daily
  Arms: Sonic-Floss toothbrush and full size brush head
Device: Routine Oral Hygiene — Oral hygiene regimen completed daily
  Arms: Manual brushing and flossing

SUMMARY:
The study is designed to evaluate the clinical changes in gingival health by measuring the reduction of gingival bleeding and inflammation over 4 weeks. Additionally, plaque removal will be evaluated after a single use (part 1) and over 4 weeks (part 2).

DETAILED DESCRIPTION:
Data will be analyzed and reported as mean. The target population is approximately 105 healthy adult volunteers. there will be three groups with 35 subjects per group. Subjects will be randomized using a simple random sample. A computer-generated randomization schedule will be prepared by the study statistician. Based on the randomization schedule, subjects will be randomly assigned in a 1:1:1 ratio.

With 35 subjects per group, the study will have 90% power to detect an average reduction in the percent of sites with BOP of 25%.

The primary outcome will be the reduction in the percentage of sites with bleeding on probing (BOP) after 4 weeks.

Reduction in the percentage of sites with BOP after 2 weeks (+/- 2 days). Reduction in the Modified Gingival index after 2 (+/- 2 days) and 4 weeks (+/- 2 days). Reduction in Rustogi Modification of Navy Plaque Index pre & Post, 2 weeks (+/- 2 days) and 4 weeks (+/- 2 days).

Data will include whole mouth, approximal, marginal, facial, and lingual analysis for all indices. Intraoral examination will be performed and any adverse events will be reported and followed-up.

Subjects will complete a questionnaure at the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Provided written informed consent prior to being entered into the study
* Have at least twenty (20) natural teeth (5 evaluable teeth in each quadrant) with scorable facial and lingual surfaces as determined by examiner
* No tobacco use or other substance via the mouth including but not limited to cigarettes, cigars, smokeless tobacco hookah, cannabis, snuff, chew, or vaping electronic cigarettes
* Have a minimum of 50% bleeding on probing sites (6 sites per tooth, total of 120 - 168 total sites)
* Have probing depths </= 4 mm
* Have a mean baseline gingival index score of >/= to 1.75 as determined by the Modified Gingival Index.
* Agree not to have a dental prophylaxis or any other elective, non-emergency dental procedures any time during the study
* Agree to abstain from the use of chewing gum, mouth rinses, any toothpaste other than the study toothpaste, tooth whitening products (either professional or at home use) and all other oral hygiene aids other than the study procedures for the duration of the study
* Agree to refrain from all oral hygiene on morning of each evaluation visit
* Agree to comply with the conditions ad schedule of the study

Exclusion Criteria:

* Physical limitations or restrictions that might preclude normal tooth brushing.
* Evidence of gross oral pathology, including widespread caries or chronic neglect, extensive restoration, pre-existing gross plaque or soft or hard tissue tumor of the oral cavity.
* Heavy supra- or subgingival calculus that might interfere with evaluations as determined by the examiner.
* Evidence of major oral hard or soft tissue lesions or trauma at the baseline visit as determined by the examiner.
* Conditions requiring antibiotic treatment prior to dental procedures.
* History of uncontrolled diabetes or hepatic or renal disease, or other serious conditions or transmittable disease, (e.g. cardiomyopathy, immunocompromised).
* Subjects with several fully crowned or extensively restored teeth, orthodontic appliances, peri/oral piercings, or removable partial dentures.
* Treatment with antibiotics within 6 months before the baseline examination, or a condition that is likely to require antibiotic treatment over the course of the trial.
* Chronic treatment (2-weeks or more) with any medication known to affect periodontal status (including phenytoin, calcium antagonists, cyclosporine, Coumadin, nonsteroidal anti-inflammatory drugs, and aspirin (325 mg)) within the month before the baseline examination. All other medications for chronic medical conditions must have been initiated at least 3 months before enrollment.
* Have severe periodontal disease or being actively treated for periodontal disease.
* Having history of early-onset periodontitis or acute necrotizing ulcerative gingivitis.
* Concomitant periodontal therapy other than prophylaxis in the last 3 months.
* Professional prophylaxis within 1 month prior to the baseline clinical evaluation.
* Subjects who participated in a gingivitis study in the past month.
* History of significant adverse event following use of oral hygiene products such as toothpastes and mouth rinses.
* Self-reported pregnancy or lactating women or planning to become pregnant during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
Bleeding on Probing | 4 weeks
  Binary measure of present = 1 or absent =0. Mean score is determined by adding the total number of sites with bleeding (six per tooth) and dividing by the total evaluable sites.
Modified Gingival Index | 4 weeks
  Index uses a 0 - 4 point scale

SECONDARY OUTCOMES:
Rustogi Modification of the Navy Plaque Index | 4 weeks
  Each tooth is scored using 9 sections for the facial and lingual surfaces.

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy G Qaqish, BSc, Study Director — All Sum Research Center Ltd.
Locations (1):
- All Sum Research Center, Mississauga, Ontario, Canada